CLINICAL TRIAL: NCT03996837
Title: Evaluation of the Application Platelet Rich Plasma in the Treatment of Patients With Recurrent Implantation Failure in IVF-ICSI & Freeze Embryo Transfer Cycles in Royan Institute; a Randomized Controlled Trial
Brief Title: Platelet Rich Plasma and Recurrent Implantation Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRP-RIF
Record Dates: First submitted 2019-05-26; First posted 2019-06-25 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Recurrent Implantation Failure
Keywords: Platelet rich plasma; Recurrent implantation failure; Infertility; Assisted reproduction technology
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fresh embryo transfer with intra uterine infusion of PRP (Experimental): In IVF-ICSI cycles, ovulation will be stimulated through the standard protocol using a gonadotropin-releasing hormone agonist for all patients. 48 hours after the oocyte retrieval and ensuring that at least 3 good quality embryos are formed, patients will be randomized into two groups of with and without PRP intrauterine injection. For all patients, 2 embryos in the blastocyst stage with excellent or good quality will be transferred. One milliliter PRP will be injected into the patients' uterine cavity using an embryo transfer catheter (Labotect Gmbh, Labor-Technik-Gottingen Kampweg 12, 37124 Rosdorf, Germany) 48 hours before embryo transfer. In order to eliminate the effects of catheter insertion, the same catheter will be applied to the patients in the control group 48 hours before the embryo transfer without any injections.
  Interventions: Other: Intra uterine infusion of platelet rich plasma
- Fresh embryo transfer without intra uterine infusion of PRP (No Intervention): In IVF-ICSI cycles, ovulation will be stimulated through the standard protocol using a gonadotropin-releasing hormone agonist for all patients. 48 hours after the oocyte retrieval and ensuring that at least 3 good quality embryos are formed, patients will be randomized into two groups of with and without PRP intrauterine injection. For all patients, 2 embryos in the blastocyst stage with excellent or good quality will be transferred. One milliliter PRP will be injected into the patients' uterine cavity using an embryo transfer catheter (Labotect Gmbh, Labor-Technik-Gottingen Kampweg 12, 37124 Rosdorf, Germany) 48 hours before embryo transfer. In order to eliminate the effects of catheter insertion, the same catheter will be applied to the patients in the control group 48 hours before the embryo transfer without any injections.
- Freeze embryo transfer with intra uterine infusion of PRP (Experimental): In frozen embryos transfer cycles, the endometrium of all patients will be prepared through the standard protocol using a gonadotropin-releasing hormone agonist. Following this process, 2 embryos in the blastocyst stage with good or excellent quality will be transferred. It is worth mentioning that in 48 hours prior to the embryo transfer; 1 mL of PRP will be injected into the uterine cavity using an embryo transfer catheter. In order to eliminate the effects of catheter insertion, the same catheter will be applied to the patients in the control group 48 hours before the embryo transfer without any injections.
  Interventions: Other: Intra uterine infusion of platelet rich plasma
- Freeze embryo transfer without intra uterine infusion of PRP (No Intervention): In frozen embryos transfer cycles, the endometrium of all patients will be prepared through the standard protocol using a gonadotropin-releasing hormone agonist. Following this process, 2 embryos in the blastocyst stage with good or excellent quality will be transferred. It is worth mentioning that in 48 hours prior to the embryo transfer; 1 mL of PRP will be injected into the uterine cavity using an embryo transfer catheter. In order to eliminate the effects of catheter insertion, the same catheter will be applied to the patients in the control group 48 hours before the embryo transfer without any injections.

INTERVENTIONS:
Other: Intra uterine infusion of platelet rich plasma — Platelet Rich Plasma (PRP) is a blood product with a high platelet and a normal plasma fibrinogen level. Given the effective factors of RPR in repairing damaged tissues, its application in the field of regenerative medicine has widely been interested over the last three decades. According to the literature, PRP is an effective and safe treatment in the fields of orthopaedics, dermatology, ophthalmology, and repair of neurological, vascular, and connective tissue damage, but its application in the field of infertility is limited to a few pilot studies in which the effects of PRP on endometrium and recurrent implantation failure (RIF) were investigated.
  Arms: Freeze embryo transfer with intra uterine infusion of PRP; Fresh embryo transfer with intra uterine infusion of PRP

SUMMARY:
This study is a randomized controlled clinical trial to compare the pregnancy outcomes of infertile women with recurrent implantation failure. The study population consisted of infertile women with a history of recurrent implantation failure who had failed to achieve a clinical pregnancy which at least four good quality embryos transfers and are now candidate for IVF-ICSI or freeze embryo transfer cycles with and without intra uterine infusion of platelet rich plasma in Reproductive Biomedicine Research Center, Royan institute, Tehran Iran.

DETAILED DESCRIPTION:
Platelet Rich Plasma (PRP) is a blood product with a high platelet and a normal plasma fibrinogen level. Given the effective factors of RPR in repairing damaged tissues, its application in the field of regenerative medicine has widely been interested over the last three decades. According to the literature, PRP is an effective and safe treatment in the fields of orthopaedics, dermatology, ophthalmology, and repair of neurological, vascular, and connective tissue damage, but its application in the field of infertility is limited to a few pilot studies in which the effects of PRP on endometrium and recurrent implantation failure (RIF) were investigated. Given the importance of endometrial compliance and according to molecular studies, which indicate that endometrial growth factors in women with a history of RIF are lower than normal fertile women, PRP, along with other existing strategies, can be used to improve endometrial compliance in patients with a history of RIF. The present randomized, controlled clinical trial is proposed to determine the efficacy of PRP in the treatment of patients with RIF in the cycles of IVF-ICSI and frozen embryo transfer at Royan Institute.

ELIGIBILITY:
Inclusion Criteria:

1. Infertile women with a history of recurrent implantation failure who had failed to achieve a clinical pregnancy which at least four good quality embryos transfers
2. 20<Age<40
3. 19<BMI<29
4. Non endocrine, hematologic and autoimmune disorders
5. Non chromosomal and genetic abnormalities
6. Non uterine anomalies, surgical history, endometriosis, adenomyosis, hydro salpinx, uterine fibroids, Polycystic ovary syndrome
7. Having at least three good quality embryos

Exclusion Criteria:

1. Cervicitis
2. Recent fever condition
3. Use of corticosteroids (in up to 2 weeks before the procedure) or non-steroid anti-inflammatories (in up to 48 hours before procedure)
4. Anemia, thrombocytopenia, platelet dysfunction syndrome, hypofibrinogenemia
5. Septicemia, active infections with Pseudomonas, Klebsiella or Enterococcus
6. History of cancer
7. Patient's tendency for withdrawal

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
Implantation rate | 4-6 weeks after embryo transfer
  The number of gestational sacs observed, divided by the number of embryos transferred

SECONDARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks after embryo transfer
  Continued pregnancy at > gestational week 12 or more per initiated cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Royan Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yahyaei A, Madani T, Vesali S, Mashayekhi M. Intrauterine infusion of autologous platelet rich plasma can be an efficient treatment for patients with unexplained recurrent implantation failure. Sci Rep. 2024 Oct 29;14(1):26009. doi: 10.1038/s41598-024-77578-1. PMID 39472511